CLINICAL TRIAL: NCT01528384
Title: A Phase 1 Study of ADI PEG 20 in Pediatric Subjects Who Are Argininosuccinate Synthetase (ASS) Deficient and Have Failed Prior Systemic Therapy
Brief Title: Ph 1 Study of ADI PEG 20 in Pediatric Subjects Who Are Argininosuccinate Synthetase (ASS) Deficient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2009-002
Record Dates: First submitted 2012-01-14; First posted 2012-02-08 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Argininosuccinate Synthetase Deficient
Keywords: Arginine; Arginine deiminase; Argininosuccinate synthetase; Phase 1; Pediatric; Failed other treatments; Pediatric patients
MeSH Terms: interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ADI-PEG 20 — 4.5, 9 and 18 mg/m2 dosage weekly dosing intramuscular until progressive disease
  Other Names: pegylated arginine deiminase

SUMMARY:
This is a phase 1 study of pegylated arginine deiminase (ADI-PEG 20) in pediatric patients who deficient in the expression of tumor argininosuccinate synthetase, and have failed prior treatments. The study hypothesis is that this drug will be safe in pediatric patients.

DETAILED DESCRIPTION:
This phase 1 study will use a classic 3 dose levels by 3 patients per dose level design. Once the maximum tolerated dose is reached, additional patients may be enrolled at that dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of failed current standard treatment(s), or AEs associated with prior systemic agent(s) that resulted in discontinuance of that agent(s).
2. Argininosuccinate synthetase deficient tumor.
3. Measurable disease as assessed by >5% blasts on bone marrow aspirate for patients with leukemia or using RECIST 1.1 criteria for solid tumors.
4. Age 4 to ≤ 18 years.
5. No prior systemic treatment for the tumor in the last 2 weeks for solid tumors and 1 week for leukemia, except hydroxyurea used only to control very high WBC.
6. Fully recovered from any prior surgery and no major surgery within 4 weeks of initiating treatment. Surgery for placement of vascular access devices is acceptable.
7. Female subjects of 10 years and older and male subjects must be asked to use appropriate contraception for both the male and female for the duration of the study.
8. No concurrent investigational studies are allowed.
9. For solid tumor subjects only: Absolute neutrophil count (ANC) >750/µL.
10. For solid tumor subjects only: Platelets >50,000/µL.
11. For solid tumor subjects only: Serum uric acid ≤ 8 mg/dL (with or without medication control).
12. Serum creatinine ≤ 1.5 x the upper limit of normal range, or, if serum creatinine >1.5 x the upper limit of normal range, then the creatinine clearance must be ≥ 60 mL/min.

Exclusion Criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness.
5. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline or ≤ Grade 1 AEs due to agents administered.
6. Subjects who had been treated with ADI-PEG 20 previously.
7. History of seizure disorder not related to underlying cancer.
8. Known HIV positivity.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in laboratory values. | 2 years
  Change from baseline in laboratory values, as a measure of safety.

SECONDARY OUTCOMES:
Results of diagnostic imaging using RECIST criteria. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Herzog, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States